CLINICAL TRIAL: NCT03505723
Title: PeriOperative ISchemic Evaluation-3 Trial
Acronym: POISE-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, P.J. Devereaux, Professor, Principal Investigator, Population Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018.02.08
Record Dates: First submitted 2018-03-16; First posted 2018-04-23 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Perioperative Bleeding; Venous Thrombosis; Arterial Thrombosis
Keywords: Noncardiac surgery; Myocardial injury; Perioperative myocardial infarction; Tranexamic Acid; Hypotension; Hypertension
MeSH Terms: conditions — Venous Thrombosis; Hypotension; Hypertension | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tranexamic Acid (TXA) (Active Comparator): Patients will receive a 1g loading dose of intravenous TXA before surgery and a 1g loading dose of intravenous TXA at the end of surgery (wound closure).
  Interventions: Drug: Tranexamic Acid
- Placebo (0.9% normal saline) (Placebo Comparator): Patients will receive a 1g loading dose of placebo (0.9% normal saline) before surgery and a 1g loading dose of placebo (0.9% normal saline) at the end of surgery (wound closure).
  Interventions: Drug: Placebo (Saline)
- Hypotension-avoidance strategy (Active Comparator): Aims to avoid hypotension before surgery (preoperative), during surgery (intraoperative) and for the first 2 days after the day of surgery (postoperative).
  Interventions: Other: Perioperative hypotension-avoidance strategy
- Perioperative hypertension-avoidance strategy (Placebo Comparator): Aims to avoid hypertension before surgery (preoperative), during surgery (intraoperative) and for the first 2 days after the day of surgery (postoperative).
  Interventions: Other: Perioperative hypertension-avoidance strategy

INTERVENTIONS:
Drug: Tranexamic Acid — Within 20 minutes preceding the anticipated skin incision, patients will receive intravenous TXA at a loading dose of 1g over 10 minutes, with a second 1g bolus given at the end of surgery when closing the wound.
  Other Names: TXA
  Arms: Tranexamic Acid (TXA)
Drug: Placebo (Saline) — Within 20 minutes preceding the anticipated skin incision, patients will receive intravenous placebo (0.9% normal saline) at a loading dose of 1g over 10 minutes, with a second 1g bolus given at the end of surgery when closing the wound.
  Other Names: saline
  Arms: Placebo (0.9% normal saline)
Other: Perioperative hypotension-avoidance strategy — Perioperative hypotension-avoidance strategy includes:
  1. Preoperative algorithm that only continues some antihypertensive medications in a stepwise manner for systolic BP ≥130 mm Hg before surgery,
  2. Intraoperative blood pressure targeting a mean arterial pressure (MAP) ≥80 mm Hg
  3. Postoperative algorithm that only continues some antihypertensive medications in a stepwise manner for systolic BP ≥130 mm Hg during the first 48 hours after surgery.
  Arms: Hypotension-avoidance strategy
Other: Perioperative hypertension-avoidance strategy — Perioperative hypertension-avoidance strategy (i.e., routine care) continues all antihypertensive drugs before and after surgery and an intraoperative BP strategy targeting a MAP ≥60 mm Hg.
  Arms: Perioperative hypertension-avoidance strategy

SUMMARY:
This study is a multicentre, international, randomized controlled trial of tranexamic acid (TXA) versus placebo and, using a partial factorial design, of a perioperative hypotension-avoidance versus hypertension-avoidance strategy.

DETAILED DESCRIPTION:
The POISE-3 study is a 10,000 patient, multicentre, international, non-inferiority randomized controlled trial of tranexamic acid (TXA) versus placebo and, using a partial factorial design, of a perioperative hypotension-avoidance versus hypertension-avoidance strategy. The primary objective of the study is to determine; if TXA is superior to placebo for the occurrence of life-threatening, major, and critical organ bleeding, and non-inferior to placebo for the occurrence of major arterial and venous thrombotic event; and to determine the impact of a hypotension-avoidance strategy versus a hypertension-avoidance strategy on the risk of vascular death and major vascular events in patients who are followed for 30 days after noncardiac surgery.

ELIGIBILITY:
Inclusion criteria:

1. Undergoing noncardiac surgery;
2. ≥ 45 years of age;
3. Expected to require at least an overnight hospital admission after surgery;
4. Provide written informed consent to participate in the POISE-3 Trial, AND
5. Fulfill ≥1 of the following 6 criteria (A-F):

A. NT-proBNP ≥200 ng/L B. History of coronary artery disease C. History of peripheral arterial disease D. History of stroke E. Undergoing major vascular surgery; OR F. Any 3 of 9 risk criteria i. Undergoing major surgery; ii. History of congestive heart failure; iii. History of a transient ischemic attack; iv. Diabetes and currently taking an oral hypoglycemic agent or insulin; v. Age >70 years; vi. History of hypertension; vii. Serum creatinine > 175 µmol/L (> 2.0 mg/dl); viii. History of smoking within 2 years of surgery; ix. Undergoing emergent/urgent surgery.

Exclusion criteria:

1. Patients undergoing cardiac surgery
2. Patients undergoing cranial neurosurgery
3. Planned use of systemic TXA during surgery
4. Low-risk surgical procedure (based on individual physician's judgment)
5. Hypersensitivity or known allergy to TXA
6. Creatinine clearance <30 mL/min (Cockcroft-Gault equation) or on chronic dialysis
7. History of seizure disorder
8. Patients with recent stroke, myocardial infarction, acute arterial thrombosis or venous thromboembolism (<3 month)
9. Patients with fibrinolytic conditions following consumption coagulopathy
10. Patients with subarachnoid hemorrhage within the past 30 days
11. Women of childbearing potential who are not taking effective contraception, pregnant or breast-feeding
12. Previously enrolled in POISE-3 Trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9535 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
A composite of life-threatening bleeding, major bleeding, and critical organ bleeding | 30 days after randomization
  Number of patients who have at least one of the following: life-threatening bleeding, major bleeding, and critical organ bleeding
A composite of MINS, non-hemorrhagic stroke, peripheral arterial thrombosis, and symptomatic proximal venous thromboembolism. | 30 days after randomization
  Number of patients who have at least one of the following: myocardial injury after noncardiac surgery, non-hemorrhagic stroke, peripheral arterial thrombosis, and symptomatic proximal venous thromboembolism.
For patients in the blood pressure management arm: A composite of vascular death, non-fatal MINS, non-fatal stroke, and non-fatal cardiac arrest. | 30 days after randomization
  Number of patients enrolled in the blood pressure management arm who have at least one of the following: vascular death, non-fatal myocardial injury after noncardiac surgery, non-fatal stroke, and non-fatal cardiac arrest.

SECONDARY OUTCOMES:
A net risk-benefit outcome as a composite of vascular death, and non-fatal life-threatening,major or critical organ bleeding,MINS,stroke,peripheral arterial thrombosis,and symptomatic proximal venous thromboembolism | 30 days after randomization
  Number of patients who have at least one of the following: vascular death, and non-fatal life-threatening, major or critical organ bleeding, myocardial injury after noncardiac surgery, stroke, peripheral arterial thrombosis, and symptomatic proximal venous thromboembolism,
BIMS | 30 days after randomization
  Number of patients who experience bleeding independently associated with mortality after noncardiac surgery (BIMS)
MINS | 30 days after randomization
  Number of patients who experience a myocardial injury after noncardiac surgery (MINS)
MINS not fulfilling the universal definition of myocardial infarction | 30 days after randomization
  Number of patients who experience a myocardial injury after noncardiac surgery (MINS) not fulfilling the 3rd universal definition of myocardial infarction
Myocardial infarction | 30 days after randomization
  Number of patients who experience a myocardial infarction
For patients in the blood pressure management arm: all-cause mortality | 30 days after randomization
  Number of patients who die of any cause
For patients in the blood pressure management arm: MINS | 30 days after randomization
  Number of patients who experience a myocardial injury after noncardiac surgery (MINS)
For patients in the blood pressure management arm: Myocardial infarction | 30 days after randomization
  Number of patients who experience a myocardial infarction
For patients in the blood pressure management arm: MINS not fulfilling the universal definition of myocardial infarction | 30 days after randomization
  Number of patients who experience MINS not fulfilling the universal definition of myocardial infarction

OTHER OUTCOMES:
Life threatening bleeding | 30 days after randomization
  Number of patients who experience a life threatening bleed.
Major bleeding | 30 days after randomization
  Number of patients who experience a major bleed.
Critical organ bleeding | 30 days after randomization
  Number of patients who experience bleeding in a critical organ.
International Society on Thrombosis and Haemostasis (ISTH) major bleeding | 30 days after randomization
  Number of patients who experience an International Society on Thrombosis and Haemostasis (ISTH) major bleeding
Non-hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a non-hemorrhagic stroke
Peripheral arterial thrombosis | 30 days after randomization
  Number of patients who experience peripheral arterial thrombosis
Symptomatic proximal venous thromboembolism | 30 days after randomization
  Number of patients who experience a symptomatic proximal venous thromboembolism
All-cause mortality | 30 days after randomization
  Number of patients who die of any cause
Vascular mortality | 30 days after randomization
  Number of patients who die of vascular cause
Hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a hemorrhagic stroke
Transfusion rate | 30 days after randomization
  Rate of transfusion in patients who experience a major bleeding event
Cardiac revascularization | 30 days after randomization
  Number of patients who have undergo cardiac revascularization
Amputation | 30 days after randomization
  Number of patients who have an amputation
Symptomatic pulmonary embolism | 30 days after randomization
  Number of patients who experience a symptomatic pulmonary embolism
Symptomatic proximal DVT | 30 days after randomization
  Number of patients who experience a symptomatic proximal DVT
Any symptomatic or asymptomatic proximal venous thromboembolism | 30 days after randomization
  Number of patients who experience any (symptomatic or asymptomatic) proximal venous thromboembolism
Acute kidney injury | 30 days after randomization
  Number of patients who experience an acute kidney injury
New renal replacement therapy | 30 days after randomization
  Number of patients who require new renal replacement therapy
Re-hospitalization for vascular reasons | 30 days after randomization
  Number of patients who experience a re-hospitalization for vascular reasons
Seizures | 30 days after randomization
  Number of patients who experience a seizure
Infection/sepsis | 30 days after randomization
  Number of patients who experience infection/sepsis
Disability | 30 days after randomization
  Number of patients who experience disability (based on 12-item WHO Disability Assessment Schedule [WHODAS 2.0]).
Length of hospital stay | 30 days after randomization
  Average length of hospital stay
Days alive and at home | 30 days after randomization
  Number of days alive and at home
For patients in the blood pressure management arm: vascular death | 30 days after randomization
  Number of patients who die from a vascular cause
For patients in the blood pressure management arm: non-fatal MINS | 30 days after randomization
  Number of patients who experience a non-fatal MINS
For patients in the blood pressure management arm: non-fatal stroke | 30 days after randomization
  Number of patients who experience a non-fatal stroke
For patients in the blood pressure management arm: non-fatal cardiac arrest | 30 days after randomization
  Number of patients who experience non-fatal cardiac arrest
For patients in the blood pressure management arm: hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a hemorrhagic stroke
For patients in the blood pressure management arm: non-hemorrhagic stroke | 30 days after randomization
  Number of patients who experience a non-hemorrhagic stroke
For patients in the blood pressure management arm: acute kidney injury | 30 days after randomization
  Number of patients who experience an acute kidney injury
For patients in the blood pressure management arm: new renal replacement therapy | 30 days after randomization
  Number of patients with new requirement for renal replacement therapy
For patients in the blood pressure management arm: acute congestive heart failure | 30 days after randomization
  Number of patients who experience acute congestive heart failure
For patients in the blood pressure management arm: new clinically important atrial fibrillation | 30 days after randomization
  Number of patients who experience new clinically important atrial fibrillation
For patients in the blood pressure management arm: sepsis | 30 days after randomization
  Number of patients who experience a sepsis event
For patients in the blood pressure management arm: disability | 30 days after randomization
  Number of patients who experience disability (based on 12-item WHO Disability Assessment Schedule [WHODAS 2.0]).
For patients in the blood pressure management arm: cancellation/postponement of surgery on the day of surgery due to BP concerns | 30 days after randomization
  Number of patients whose surgery was cancelled/postponed on the day of surgery due to BP concerns
For patients in the blood pressure management arm: length of hospital stay | 30 days after randomization
  Average length of hospital stay required
For patients in the blood pressure management arm: days alive and at home | 30 days after randomization
  Number of days alive and at home
All-cause mortality | 1 year after randomization
  Number of patients who die of any cause
Vascular mortality | 1 year after randomization
  Number of patients who die of vascular cause
Myocardial infarction | 1 year after randomization
  Number of patients who experience a myocardial infarction
Cardiac arrest | 1 year after randomization
  Number of patients who experience cardiac arrest
Hemorrhagic stroke | 1 year after randomization
  Number of patients who experience a hemorrhagic stroke
Non-hemorrhagic stroke | 1 year after randomization
  Number of patients who experience a non-hemorrhagic stroke
Peripheral arterial thrombosis | 1 year after randomization
  Number of patients who experience peripheral arterial thrombosis
Amputation | 1 year after randomization
  Number of patients who had an amputation
Symptomatic pulmonary embolism | 1 year after randomization
  Number of patients who experience a symptomatic pulmonary embolism
Symptomatic proximal DVT | 1 year after randomization
  Number of patients who experience a symptomatic proximal DVT
Symptomatic proximal venous thromboembolism | 1 year after randomization
  Number of patients who experience a symptomatic proximal venous thromboembolism
Any symptomatic or asymptomatic proximal venous thromboembolism | 1 year after randomization
  Number of patients who experience any symptomatic or asymptomatic proximal venous thromboembolism
New renal replacement therapy | 1 year after randomization
  Number of patients who require new renal replacement therapy
Re-hospitalization for vascular reasons | 1 year after randomization
  Number of patients re-hospitalized for vascular reasons
Seizures | 1 year after randomization
  Number of patients who experience a seizure
Infection/sepsis | 1 year after randomization
  Number of patients who experience an infection and/or sepsis event
Disability | 1 year after randomization
  Number of patients who experience disability (based on 12-item WHO Disability Assessment Schedule [WHODAS 2.0]).
For patients in the blood pressure management arm: all-cause mortality | 1 year after randomization
  Number of patients who die of any cause
For patients in the blood pressure management arm: vascular mortality | 1 year after randomization
  Number of patients who die of a vascular cause
For patients in the blood pressure management arm: myocardial infarction | 1 year after randomization
  Number of patients who experience a myocardial infarction
For patients in the blood pressure management arm: cardiac arrest | 1 year after randomization
  Number of patients who experience cardiac arrest
For patients in the blood pressure management arm: hemorrhagic stroke | 1 year after randomization
  Number of patients who experience a hemorrhagic stroke
For patients in the blood pressure management arm: non-hemorrhagic stroke | 1 year after randomization
  Number of patients who experience a non-hemorrhagic stroke
For patients in the blood pressure management arm: new renal replacement therapy | 1 year after randomization
  Number of patients who require new renal replacement therapy
For patients in the blood pressure management arm: acute congestive heart failure | 1 year after randomization
  Number of patients who experience acute congestive heart failure
For patients in the blood pressure management arm: sepsis | 1 year after randomization
  Number of patients who experience a sepsis event
For patients in the blood pressure management arm: Disability | 1 year after randomization
  Number of patients who experience disability (based on 12-item WHO Disability Assessment Schedule [WHODAS 2.0]).
For patients in the blood pressure management arm (CogPOISE-3 Sub study): Delirium | Post operative day one to three
  Number of patients who experience delirium (based on 3D-CAM or ICU-CAM)
For patients in the blood pressure management arm (CogPOISE-3 Sub study): Cognitive decline | 1 year after randomization
  Number of patients who experience cognitive decline (at least 2 points decline on Montreal Cognitive Assessment MoCA) compared to assessment after consent and before randomization

CONTACTS AND LOCATIONS:
Overall Officials: PJ Devereaux, MD, PhD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (114):
- United States (12):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Cleveland Clinic, Florida, Weston, Florida
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Cleveland Clinic - Fairview, Cleveland, Ohio
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Cleveland Clinic - Hillcrest, Mayfield Heights, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
- Australia (17):
  - Queen Elizabeth II Jubilee Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
  - Dandenong Hospital, Dandenong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Western Health, Footscray
  - Peter MacCallum Hospital, Melbourne
  - John Hunter Hospital, New Lambton
  - Royal Perth, Perth
  - Princes of Wales Hospital, Randwick
  - Goulburn Valley Health, Shepparton
  - Westmead Hospital, Sydney
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - CHU Brugmann, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Brazil (2):
  - Hospital do Coracao de Pocos de Caldas, Poços de Caldas, Minas Gerais
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
- Canada (12):
  - University of Calgary, O'Brien Institute for Public Health, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital & Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - University Health Network (Toronto General Hospital), Toronto, Ontario
  - CHUM, Montreal, Quebec
  - Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital (Saskatoon), Saskatoon, Saskatchewan
  - Victoria Hospital, London
- Chile (2):
  - Clinica Santa Maria, Santiago
  - Hospital Hernan Henriquez, Temuco
- China (4):
  - Second Hospital of Anhui Medical University, Hefei, Anhui
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - West China Hospital of Sichuan University, Chengdu, Sichuan
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen, Capital Region
  - Rigshospitalet, Abdominal Centre, Copenhagen
  - Zealand University Hospital, Køge
- Groupe Hospitalier Paris Saint Joseph, Paris, France
- Germany (4):
  - University Hospital RWTH Aachen, Aachen
  - University Hospital Bonn, Bonn
  - Klinikum Dortmund gGmbH, Dortmund
  - University Hospital Düsseldorf, Düsseldorf
- Prince of Wales Hospital, Shatin, Hong Kong
- India (13):
  - Surat Institute of Digestive Science, Surat, Gujarat
  - Sumandeep Vidyapeeth & Dhiraj General Hospital, Vadodara, Gujurat
  - Nanjappa Hospital, Shimoga, Karnataka
  - Government Medical College, Trivandrum, Kerala
  - Rahate Surgical Hospital, Nagpur, Maharashtra
  - Sengupta Hospital & Research Institute, Nagpur, Maharashtra
  - AMAI Charitable Trust's Ace Hospital, Pune, Maharashtra
  - Sidhu Hospital Pvt. Ltd., Dorāha, Punjab
  - Christian Medical College, Ludhiana, Ludhiana, Punjab
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Lucknow, Uttar Pradesh
  - NH Rabindranath Tagore International Inst. of Cardiac Sciences, Kolkata, West Bengal
  - TD Medical College, Alappuzha
  - Bangalore Baptist Hospital, Bangalore
- Italy (4):
  - Ospedale Galliera di Genova, Genova
  - Instituto Clinico San Siro, Milan
  - IRCCS San Raffaele Scientific Institute, Milan
  - IRCCS Galeazzi Orthopedic Institute, Milan
- Malaysia (6):
  - Port Dickson Hospital, Port Dickson, Negeri Sembilan
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Pulau Pinang, Pulau Pinang
  - Sungai Buloh Hospital, Sungai Buloh
- Netherlands (2):
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Erasmus University Medical Center, Rotterdam
- New Zealand (3):
  - Auckland General Hospital, Grafton, Auckland
  - Middlemore Hospital, Auckland
  - Waikato District Health Board, Hamilton
- Pakistan (2):
  - Shifa International Hospitals, Islamabad, Islamabad
  - Aga Khan University, Karachi
- Poland (3):
  - Jagiellonian University Medical College, Krakow
  - Specialistyczny Szpital im. E. Szczeklika w Tarnowie, Tarnów
  - Szpital Uniwersytecki im Karola Marcinkowskiego w Zielonej Górze, Zielona Góra
- Russia (7):
  - City Hospital 1 of Arkhangelsk, Arkhangelsk
  - V. Negovskiy Reanimatology Research Institute, Moscow
  - Moscow Regional Research & Clinical Institute (MONIKI), Moscow
  - City Hospital N25, Novosibirsk
  - E. Meshalkin National Medical Research Center, Novosibirsk
  - Hospital of Saint-Petersburg State University, Saint Petersburg
  - Tyumen State Medical University, Tyumen
- South Africa (3):
  - Groote Schuur Hospital, Observatory, Cape Town
  - Sefako Makgatho Health Sciences University (SMU), Ga-Rankuwa, Gauteng
  - Steve Biko Academic Hospital - University of Pretoria, Pretoria, Gauteng
- Spain (7):
  - Hospital Clinic - Barcelona, Barcelona
  - Hospital de la Sta Creu i Sant Pau, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital Clínico Universitario in Valladolid, Valladolid
- United Kingdom (3):
  - Medway NHS Foundation Trust, Gillingham
  - Chelsea & Westminster Hospital, London
  - West Middlesex Hospital, London

REFERENCES:
- [Derived] Marcucci M, Chan MTV, Painter TW, Efremov S, Aguado HJ, Astrakov SV, Kleinlugtenbelt YV, Patel A, Cata JP, Amir M, Kirov M, Leslie K, Duceppe E, Borges FK, de Nadal M, Tandon V, Landoni G, Likhvantsev VV, Lomivorotov V, Sessler DI, Martinez-Zapata MJ, Xavier D, Fleischmann E, Wang CY, Meyhoff CS, Wittmann M, Torres D, Highton D, Jacka M, B V, Zarnke K, Sidhu RS, Oriani G, Ayad S, Minear S, Weaver TE, Ruetzler K, Brusasco C, Parlow JL, Maxwell E, Miller S, Mrkobrada M, Bhatt KSC, Rahate P, Kowark A, De Blasio G, Ofori SN, Conen D, Srinathan S, Szczeklik W, Jayaram R, Ellerkmann RK, Momeni M, Copland I, Vincent J, Balasubramanian K, Li Z, Wang MK, Li D, McGillion MH, Kurz A, Sharma M, Short TG, Devereaux PJ; cogPOISE-3 Trial Investigators and Study Groups. Effects of a Hypotension-Avoidance Versus a Hypertension-Avoidance Strategy on Neurocognitive Outcomes After Noncardiac Surgery. Ann Intern Med. 2025 Jul;178(7):909-920. doi: 10.7326/ANNALS-24-02841. Epub 2025 Jun 3. PMID 40456161
- [Derived] Park LJ, Marcucci M, Ofori SN, Borges FK, Nenshi R, Kanstrup CTB, Rosen M, Landoni G, Lomivorotov V, Painter TW, Xavier D, Martinez-Zapata MJ, Szczeklik W, Meyhoff CS, Chan MTV, Simunovic M, Bogach J, Serrano PE, Balasubramanian K, Cadeddu M, Yang I, Kim WH, Devereaux PJ. Safety and Efficacy of Tranexamic Acid in General Surgery. JAMA Surg. 2025 Mar 1;160(3):267-274. doi: 10.1001/jamasurg.2024.6048. PMID 39813061
- [Derived] POISE-3 Trial Investigators and Study Groups. A sub-study of the POISE-3 randomized trial examined effects of a perioperative hypotension-avoidance strategy versus a hypertension-avoidance strategy on the risk of acute kidney injury. Kidney Int. 2025 Jan;107(1):155-168. doi: 10.1016/j.kint.2024.10.007. Epub 2024 Oct 25. PMID 39490985
- [Derived] Marcucci M, Painter TW, Conen D, Lomivorotov V, Sessler DI, Chan MTV, Borges FK, Leslie K, Duceppe E, Martinez-Zapata MJ, Wang CY, Xavier D, Ofori SN, Wang MK, Efremov S, Landoni G, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Ruetzler K, Parlow JL, Tandon V, Fleischmann E, Polanczyk CA, Lamy A, Jayaram R, Astrakov SV, Wu WKK, Cheong CC, Ayad S, Kirov M, de Nadal M, Likhvantsev VV, Paniagua P, Aguado HJ, Maheshwari K, Whitlock RP, McGillion MH, Vincent J, Copland I, Balasubramanian K, Biccard BM, Srinathan S, Ismoilov S, Pettit S, Stillo D, Kurz A, Belley-Cote EP, Spence J, McIntyre WF, Bangdiwala SI, Guyatt G, Yusuf S, Devereaux PJ; POISE-3 Trial Investigators and Study Groups. Hypotension-Avoidance Versus Hypertension-Avoidance Strategies in Noncardiac Surgery : An International Randomized Controlled Trial. Ann Intern Med. 2023 May;176(5):605-614. doi: 10.7326/M22-3157. Epub 2023 Apr 25. PMID 37094336
- [Derived] Devereaux PJ, Marcucci M, Painter TW, Conen D, Lomivorotov V, Sessler DI, Chan MTV, Borges FK, Martinez-Zapata MJ, Wang CY, Xavier D, Ofori SN, Wang MK, Efremov S, Landoni G, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Duceppe E, Ruetzler K, Parlow JL, Tandon V, Fleischmann E, Polanczyk CA, Lamy A, Astrakov SV, Rao M, Wu WKK, Bhatt K, de Nadal M, Likhvantsev VV, Paniagua P, Aguado HJ, Whitlock RP, McGillion MH, Prystajecky M, Vincent J, Eikelboom J, Copland I, Balasubramanian K, Turan A, Bangdiwala SI, Stillo D, Gross PL, Cafaro T, Alfonsi P, Roshanov PS, Belley-Cote EP, Spence J, Richards T, VanHelder T, McIntyre W, Guyatt G, Yusuf S, Leslie K; POISE-3 Investigators. Tranexamic Acid in Patients Undergoing Noncardiac Surgery. N Engl J Med. 2022 May 26;386(21):1986-1997. doi: 10.1056/NEJMoa2201171. Epub 2022 Apr 2. PMID 35363452
- [Derived] Marcucci M, Painter TW, Conen D, Leslie K, Lomivorotov VV, Sessler D, Chan MTV, Borges FK, Martinez Zapata MJ, Wang CY, Xavier D, Ofori SN, Landoni G, Efremov S, Kleinlugtenbelt YV, Szczeklik W, Schmartz D, Garg AX, Short TG, Wittmann M, Meyhoff CS, Amir M, Torres D, Patel A, Duceppe E, Ruetzler K, Parlow JL, Tandon V, Wang MK, Fleischmann E, Polanczyk CA, Jayaram R, Astrakov SV, Rao M, VanHelder T, Wu WKK, Cheong CC, Ayad S, Abubakirov M, Kirov M, Bhatt K, de Nadal M, Likhvantsev V, Iglesisas PP, Aguado HJ, McGillion M, Lamy A, Whitlock RP, Roshanov P, Stillo D, Copland I, Vincent J, Balasubramanian K, Bangdiwala SI, Biccard B, Kurz A, Srinathan S, Petit S, Eikelboom J, Richards T, Gross PL, Alfonsi P, Guyatt G, Belley-Cote E, Spence J, McIntyre W, Yusuf S, Devereaux PJ. Rationale and design of the PeriOperative ISchemic Evaluation-3 (POISE-3): a randomized controlled trial evaluating tranexamic acid and a strategy to minimize hypotension in noncardiac surgery. Trials. 2022 Jan 31;23(1):101. doi: 10.1186/s13063-021-05992-1. PMID 35101083